CLINICAL TRIAL: NCT03672318
Title: Phase I Study of Autologous CAR T-Cells Targeting the CD138 Antigen for Relapsed or Refractory Multiple Myeloma
Brief Title: Study of ATLCAR.CD138 Cells for Relapsed/Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1603-ATL
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Immune System Diseases
Keywords: CAR T cells; CD138; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAR138 T cells (Experimental): The first 3 subjects enrolled in the study will receive 5x10^6 CAR138 T-cells/m^2 via infusion. The number of cells for the infusion will be increased to 1x10^7 CAR138 T-cells/m^2 and then, 2.5x10^7 CAR138 T-cells/m^2, 5x10^7 CAR138 T-cells/m^2, 1x10^8 CAR138 T-cells/m^2 and 2x10^8 CAR138 T-cells/m^2 in subsequent cohorts of 3 subjects provided no dose limiting toxicities (DLTs) are observed within 4 weeks of the cell infusion. Cohort enrollment will be staggered, requiring each subject to complete at least 2 weeks of safety monitoring following CAR138 T-cell infusion at the designated dose level for the cohort before another subject is allowed to enroll in the cohort.
  Interventions: Drug: CAR138 T Cells

INTERVENTIONS:
Drug: CAR138 T Cells — The MTD is defined as the dose at which approximately 0.20 of subjects experience DLT dose escalation guided by the continual reassessment method (CRM).
  Six dose levels will be evaluated:
  Dose level 1: 5X10^6 cells/m^2 Dose level 2: 1X10^7 cells/m^2 Dose level 3: 2.5X10^7 cells/m^2 Dose level 4: 5X10^7 cells/m^2 Dose level 5: 1x10^8 cells/m^2 Dose level 6: 2x10^8 cells/m^2
  Six subjects will be enrolled at the MTD to better characterize safety at that dose level.
  Cell Administration: CAR138 T cells will be given by intravenous injection over through either a peripheral or a central line.
  The lymphodepletion regimen will consist of intravenous cyclophosphamide 300 mg/m^2 and fludarabine 30 mg/m^2 given once daily for three days.
  Other Names: ATLCAR.CD138; CAR.CD138 T cells

SUMMARY:
The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are proteins that protect the body from disease caused by bacteria or toxic substances. Antibodies work by binding those bacteria or substances, which stops them from growing and causing bad effects. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected. Both antibodies and T cells have been used to treat subjects with cancers. They both have shown promise, but neither alone has been sufficient to cure most subjects. This study is designed to combine both T cells and antibodies to create a more effective treatment. The treatment that is being researched is called autologous T lymphocyte chimeric antigen receptor cells targeted against the CD138 antigen (CAR138 T cells).

In previous studies, it has been shown that a new gene can be put into T cells that will increase their ability to recognize and kill cancer cells. A gene is a unit of DNA. Genes make up the chemical structure carrying the subject's genetic information that may determine human characteristics (i.e., eye color, height and sex). The new gene that is put in the T cells in this study makes a piece of an antibody called anti-CD138. This antibody floats around in the blood and can detect and stick to cancer cells called multiple myeloma cells because they have a substance on the outside of the cells called CD138. Anti-CD138 antibodies have been used to treat people with multiple myeloma, but have not been strong enough to cure most subjects. For this study, the anti-CD138 antibody has been changed so that instead of floating free in the blood part of it is now joined to the T cells. Only the part of the antibody that sticks to the multiple myeloma cells is attached to the T cells instead of the entire antibody. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD138 chimeric (combination) receptor-activated T cells seem to kill some of the tumor, but they do not last very long in the body and so their chances of fighting the cancer are unknown.

DETAILED DESCRIPTION:
Cell Procurement Up to 300 mL total of peripheral blood (up to 3 collections) will be obtained from subjects for cell procurement. In subjects with a low CD3 count in the peripheral blood (less than 200/μl by flow cytometry), a leukopheresis may be performed to isolate sufficient T-cells. The parameters for pheresis will be 2 blood volumes.

CAR138 T-cell Administration Autologous CAR138 T-cells will be administered 2-14 days following lymphodepletion. The lymphodepletion regimen will consist of Cyclophosphamide 300 mg/m^2 and Fludarabine 30 mg/m^2 IV each given daily over 3 consecutive days.

Duration of Therapy Autologous CAR138 T-cells will be administered 2-14 days following lymphodepletion with cyclophosphamide and fludarabine by a licensed provider (oncology registered nurse or physician) via intravenous injection over 5-10 minutes through either a peripheral or central line. The expected volume is 1-50cc.

Treatment with one infusion will be administered unless:

* The subject decides to withdraw from the study, OR
* General or specific changes in the subject's condition render the subject unacceptable for further treatment in the judgment of the investigator.

Duration of Follow-up Subjects will be followed for up to 15 years for replication-competent retrovirus evaluation or until death, whichever occurs first. Subjects removed from study for unacceptable adverse events will continue follow up for evaluation of progression free survival, overall survival and replication-competent retrovirus monitoring.

Subjects who experience disease progression after receiving a cell infusion will still be required to complete abbreviated follow up procedures.

Arms and Interventional ArmTitle : CAR138 T cells Description: The first 3 subjects enrolled in the study will receive 5x10^6 CAR138 T-cells/m^2 via infusion. The number of cells for the infusion will be increased to 1x10^7 CAR138 T-cells/m^2 and then, 2.5x10^7 CAR138 T-cells/m^2, 5x10^7 CAR138 T-cells/m^2, 1x10^8 CAR138 T-cells/m^2 and 2x10^8 CAR138 T-cells/m^2 in subsequent cohorts of 3 subjects provided no dose limiting toxicities (DLTs) are observed within 4 weeks of the cell infusion. Cohort enrollment will be staggered, requiring each subject to complete at least 2 weeks of safety monitoring following CAR138 T-cell infusion at the designated dose level for the cohort before another subject is allowed to enroll in the cohort.

ELIGIBILITY:
Eligibility criteria are divided into 3 sections: 1) eligibility criteria to be fulfilled prior to cell procurement, 2) Eligibility criteria to be met prior to lymphodepletion and 3) Eligibility criteria to be met prior to CAR138 T cell infusion.

Note: During the period of cell procurement and CAR138 T-cell production, subjects are allowed to receive additional standard of care chemotherapy or radiation therapy to stabilize their multiple myeloma if the treating physician feels it is in the subject's best interests. For subjects requiring bridging chemotherapy and/or radiation therapy while awaiting manufacture of their CAR138-T cells, details regarding treatment(s) administered including doses, frequency, number of cycles, etc. will be collected.

1. Eligibility criteria to be fulfilled prior to cell procurement

   Subjects must fulfill all of the following criteria to participate in this study.

   Written informed consent and HIPAA authorization for release of personal health information. Subjects must sign a consent to undergo cell procurement.

   Age ≥ 18 years at the time of consent.

   Karnofsky score of ≥ 60%.

   Diagnosis of relapsed or refractory multiple myeloma (as defined by the Revised Uniform Response Criteria outlined by the IMWG

   Measurable disease as defined by one or more of the following: 1) serum M-protein

   ≥1.0 g/dL (≥0.5 g/dL for IgA myeloma); 2) urine M-protein ≥200 mg/24 hours; 3) involved serum free light chain level ≥10 mg/dL AND an abnormal serum free light chain ratio. Subjects with non-secretory disease and a baseline marrow burden of myeloma of at least 30% will also be eligible to participate.

   Received at least 3 lines of prior chemotherapy. The prior regimens must have included an immunomodulatory agent (lenalidomide or pomalidomide) and a proteasome inhibitor (bortezomib, carfilzomib or ixazomib).
   * Two lines of therapy will be allowed if the subject has disease that is refractory to both an immunomodulatory agent (lenalidomide or pomalidomide) and a proteasome inhibitor.

   Received high dose melphalan followed by autologous stem-cell transplant (ASCT) or is not eligible for or has declined the procedure.

   Allogeneic stem cell transplantation is allowed provided the subject is ≥ 1 year from immunosuppressive therapy to treat/prevent graft-versus-host disease, has no evidence of active graft-versus-host disease, and has no evidence of active infection.

   Women of childbearing potential (WOCBP) should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study (starting prior to procurement), and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The male partner of WOCBP subjects enrolled into the trial should use a condom and female participants must take the responsibility to inform their partners of the need to use a condom.

   Not pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).

   No tumor in a location where enlargement could cause airway obstruction.

   No diagnosis of any of the following conditions: amyloidosis, POEMS syndrome or multiple myeloma with CNS involvement.
   * Subjects with plasma cell leukemia are allowed to participate.

   No active inflammatory or infectious gastrointestinal disorder (e.g. infectious colitis, diverticulitis or inflammatory bowel disease).

   No psychiatric illness which would prevent the subject from giving informed consent, or neurological illness that the clinician believes would complicate monitoring for CNS neurotoxicity following CAR-T infusion.

   Subjects are willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.

   No medical condition, which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the subject.

   No other prior or concomitant malignancies with the exception of:
   * Non-melanoma skin cancer
   * In-situ malignancy
   * Low-risk prostate cancer after curative therapy
   * Other cancer for which the subject has been disease free for ≥ 3 years.

   Adequate cardiac function, defined as:
   * No ECG evidence of acute ischemia
   * No ECG evidence of active, clinically significant conduction system abnormalities
   * Prior to study entry, any ECG abnormality at screening not felt to put the subject at risk has to be documented by the investigator as not medically significant
   * No uncontrolled angina or severe ventricular arrhythmias
   * No clinically significant pericardial disease
   * No history of myocardial infarction within the last 6 months prior to registration
   * No Class 3 or higher New York Heart Association Congestive Heart Failure

   No active infection (fungal, bacterial or viral) including HIV, HTLV, HBV, HCV (tests can be pending at the time of cell procurement; only those samples confirming lack of active infection will be used to generate transduced cells). Note: To meet eligibility, subjects are required to be negative for HIV antibody or HIV viral load, negative for HTLV1 and 2 antibody or PCR negative for HTLV1 and 2, negative for Hepatitis B surface antigen, and negative for HCV antibody or HCV viral load.

   Demonstrate adequate organ function prior to cell procurement as defined below:
   * Creatinine Clearance using the Cockcroft-Gault formula: ≥ 50 mL/min within 60 days of cells procurement, must be ≥ 30 mL/min within 24 hours of procurement.
   * Bilirubin: ≤ 1.5 × upper limit of normal (ULN) unless attributed to Gilbert's syndrome
   * Aspartate aminotransferase (AST): ≤ 2.5 × ULN
   * Alanine aminotransferase (ALT): ≤ 2.5 × ULN
   * Oxygen saturation: ≥ 92% on room air
   * Ejection fraction: ≥ 45%
   * Platelets: ≥ 50,000 /mm^3; mm3 within 60 days of cell procurement, must be ≥ 20,000/mm3 within 24 hours of procurement.
   * ANC: ≥ 1000 /mm^3; within 60 days of cell procurement, must be ≥ 500/mm3 (0.5 × 109/L) within 24 hours of procurement.

   Negative serum pregnancy test within 72 hours prior to cell procurement for female participants of childbearing potential. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.

   Subjects who have received prior CAR-T must be ≥9 months out from prior CAR-T and have no available or more suitable treatment options in the opinion of the treating investigator than this protocol.
2. Eligibility Criteria to be fulfilled prior to lymphodepletion

   __________________________________________________ Written informed consent to enroll in the CAR T-cell therapy trial must be obtained prior to lymphodepletion.

   Karnofsky score of ≥ 60%.

   Women of childbearing potential (WOCBP) should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study (starting prior to procurement), and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The male partner of WOCBP subjects enrolled into the trial should use a condom and female participants must take the responsibility to inform their partners of the need to use a condom.

   Not pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).

   No tumor in a location where enlargement could cause airway obstruction.

   No diagnosis of any of the following conditions: amyloidosis, POEMS syndrome or multiple myeloma with CNS involvement.
   * Subjects with plasma cell leukemia are allowed to participate.

   No active inflammatory or infectious gastrointestinal disorder (e.g. infectious colitis, diverticulitis or inflammatory bowel disease).

   No psychiatric illness which would prevent the subject from giving informed consent or neurological illness that clinician believes would complicate monitoring for CNS neurotoxicity following CAR-T infusion

   Subjects are willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.

   No medical condition, which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the subject.

   No other prior or concurrent malignancies with the exception of subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial at the investigator's discretion.

   Adequate cardiac function is defined as:
   * No ECG evidence of acute ischemia
   * No ECG evidence of active, clinically significant conduction system abnormalities
   * Prior to study entry, any ECG abnormality at screening not felt to put the subject at risk has to be documented by the investigator as not medically significant
   * No uncontrolled angina or severe ventricular arrhythmias
   * No clinically significant pericardial disease
   * No history of myocardial infarction within the last 6 months prior to registration
   * No Class 3 or higher New York Heart Association Congestive Heart Failure

   No active infection (fungal, bacterial or viral) including HIV, HBV , or HCV (tests can be pending at the time of cell procurement; only those samples confirming lack of active infection will be used to generate transduced cells). Note: To meet eligibility, subjects are required to be negative for HIV antibody or HIV viral load, negative for Hepatitis B surface antigen, and negative for HCV antibody or HCV viral load.

   Subjects must have autologous transduced activated CAR138 T-cells that meet the Certificate of Analysis (CofA) acceptance criteria.

   Subjects must have stopped taking corticosteroids for at least 48 hours prior to lymphodepleting chemotherapy; No current use of systemic corticosteroids at doses ≥10mg prednisone daily or its equivalent (those receiving <10mg/day prednisone equivalent may be enrolled at discretion of the Investigator)

   Subjects must have stopped systemic chemotherapy for at least 14 days prior to lymphodepletion

   Subjects must have stopped radiation therapy for at least 7 days prior to lymphodepletion

   Subjects should have repeated multiple myeloma serologies performed within 7 days of lymphodepletion. If markers of measurable disease no longer fall within the guidelines outlined above (procurement eligibility criterion #5), the Principal Investigator should be contacted. In such an event, the subject may be allowed to receive lymphodepletion and CAR138 T-cell infusion if it is felt to be in the subject's best interests. The subject would not be evaluable for response (disease not measurable) but would be evaluable for all other safety and efficacy measures.

   Subjects must demonstrate adequate organ function prior to lymphodepletion as defined below; all tests must be obtained within 72 hours prior to lymphodepletion.
   * Absolute Neutrophil Count (ANC): ≥ 1000 cells/mm^3; subjects should not have received G-CSF or GM-CSF within 1 week or pegylated G-CSF (Neulasta) within 2 weeks of screening for lymphodepletion
   * Platelets: ≥ 50,000 cells/mm^3; subjects should not have received platelet transfusion within 1 week of screening for lymphodepletion
   * Calculated creatinine clearance: ≥ 30 mL/min using the Cockcroft-Gault formula
   * Bilirubin: ≤ 1.5 × upper limit of normal (ULN) unless attributed to Gilbert's syndrome
   * Aspartate aminotransferase (AST): ≤ AST ≤ 2.5 × ULN
   * Alanine aminotransferase (ALT): ≤ AST ≤ 2.5 × ULN
   * Pulse oximetry: ≥90% on room air

   Has not received treatment with any investigational drug within 21 days or any tumor vaccines within the previous six weeks prior to lymphodepletion.

   No major surgery within 28 days prior to lymphodepletion.

   Male subjects with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) prior to lymphodepletion through 3 months after the last dose of study therapy.

   Negative serum pregnancy test within 72 hours prior to lymphodepleting therapy for female participants of childbearing potential. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
3. Eligibility Criteria to be fulfilled prior to CAR138 T-cell infusion _______________________________________________________ Karnofsky score of ≥ 60%.

Women of childbearing potential (WOCBP) should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study (starting prior to procurement), and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The male partner of WOCBP subjects enrolled into the trial should use a condom and female participants must take the responsibility to inform their partners of the need to use a condom.

No tumor in a location where enlargement could cause airway obstruction.

The subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.

No medical condition which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the subject.

Adequate cardiac function, defined as:

* No ECG evidence of acute ischemia
* No ECG evidence of active, clinically significant conduction system abnormalities
* Prior to study entry, any ECG abnormality at screening not felt to put the subject at risk has to be documented by the Investigator as not clinically significant
* No uncontrolled angina or severe ventricular arrhythmias
* No clinically significant pericardial disease
* No history of myocardial infarction within the last 6 months prior to registration
* No Class 3 or higher New York Heart Association Congestive Heart Failure

No active infection (fungal, bacterial, or viral)

No neurological illness that the clinician believes would complicate monitoring for CNS neurotoxicity following CAR-T infusion

Evidence of adequate organ function as defined by:

* Bilirubin ≤1.5 times the upper limit of normal (ULN) unless attributed to Gilbert's Syndrome
* AST ≤ 5 times ULN
* ALT ≤ 5 times ULN
* Serum creatinine ≤1.5 time ULN
* Pulse oximetry of > 90% on room air

No current use of systemic corticosteroids at doses ≥10mg prednisone daily or its equivalent; those receiving <10mg daily may be enrolled at the discretion of the Investigator.

The subject is a good candidate for treatment with CAR138 T-cells.

Subject has no clinical indication of rapidly progressing disease in the opinion of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2039-08-18 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with dose limiting toxicities as a measure of maximum tolerated dose of CAR138 T cells | 4 weeks from infusion of the CAR138 T cells
  The maximum tolerated dose will be determined through assessment of dose limiting toxicity (DLT) experienced during the safety evaluation period. Severity and categorization of adverse events will be determined in accordance with the National Cancer Institute's Common Terminology for Adverse Events (CTCAE, version 5.0). A DLT is defined as any of the following that may, after consultation with the FDA, be considered possibly, probably, or definitely related to the study cellular products: Grade 3 and 4 cytokine release syndrome (CRS) that persists beyond 72 hours, or any Grade 5 CRS event; Grade 4 neutropenia or thrombocytopenia lasting more than 28 days from the time of CAR138 T-cell infusion. Any other ≥ Grade 3 non- hematologic toxicity (exceptions include: alopecia; grade 3 electrolyte abnormalities, hyperglycemia, diarrhea, or nausea and vomiting that can be managed with supportive care and do not persist as Grade 3 toxicities for > 72 hours)).

SECONDARY OUTCOMES:
Survival of CAR138 T cells in vivo as assessed by PCR and flow cytometry | 15 years
  Persistence of CAR138 T-cells in vivo determined by quantitative polymerase chain reaction (PCR) and flow cytometry in samples of peripheral blood.
Overall survival after infusion of CAR138 T cells | 15 years
  To determine the overall survival (OS) after infusion of CAR138 T cells in subjects with relapsed or refractory multiple myeloma. OS will be measured from the date of administration of CAR138 T-cells to the date of death.
Progression free survival after infusion of CAR138 T cells | 15 years
  Progression Free Survival (PFS) is the time from infusion of CAR138 T cells to progression or death from any cause. Subjects not known to have progressed or died at last follow-up are censored on the date of last contact. Revised Uniform Response Criteria by the International Myeloma Working Group defines progression as: Increase of 25% from lowest response value in: Serum M component with absolute increase (AI) ≥0.5 g/dL; serum M component increase ≥1 g/dL if starting M component is ≥5 g/dL and/or; Urine M component (AI ≥200 mg/24 h) and/or; in subjects without measurable serum & urine M-protein levels: difference between involved & uninvolved FLC levels (AI > 10 mg/dL); in subjects without measurable serum & urine M-protein levels, without measurable disease by FLC level, bone marrow; Development of new or definite increase in size of existing bone lesions or soft tissue plasmacytoma; Development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Overall response rate (ORR) as defined as the percentage of subjects achieving a confirmed partial response or better based on the International Myeloma Working Group (IMWG) response criteria. | 15 years
  ORR, percentage of subjects achieving a partial response or better: Complete response (CR) is Negative immunofixation of serum and urine, disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM); stringent complete response (sCR) CR plus normal FLC ratio and absence of clonal plasma cells; Immunophenotypic CR- sCR plus absence of phenotypically aberrant plasma cells in BM with minimum of 1 million total BM cells; Molecular CR -CR plus negative allele-specific oligonucleotide polymerase chain reaction. Very good partial response -Serum and urine M component detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h; Partial response ≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200 mg per 24 hr; no known evidence of progressive or new bone lesions if radiographic studies were performed.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Tuchman, MD, MHS, Principal Investigator — Assoc. Professor, Dir. of the UNC MM and Amyloidosis Program, UNC LCCC
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trial — http://unclineberger.org/patientcare/clinical-trials/clinical-trials